CLINICAL TRIAL: NCT01419275
Title: Quantifying Collateral Perfusion in Cerebrovascular Disease-Moyamoya Disease and Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Greg Zaharchuk, Principle Investigator, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-06152011-7929
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Cerebrovascular Accident; Moyamoya Disease
MeSH Terms: conditions — Stroke; Moyamoya Disease | interventions — Magnetic Resonance Imaging

ARMS (4):
- Moyamoya (Experimental): Approximately 60 Moyamoya patients will be enrolled, and will receive arterial spin label MRI with Xenon contrast agent to assess collateral blood flow.
  Interventions: Drug: Xenon contrast agent; Device: Magnetic Resonance Imaging
- Acute stroke (Experimental): Approximately 60 acute stroke patients will be enrolled, and will receive arterial spin label MRI with Xenon contrast agent to assess collateral blood flow.
  Interventions: Drug: Xenon contrast agent; Device: Magnetic Resonance Imaging
- Healthy participants (Experimental): Approximately 30 healthy participants will be enrolled, and will receive arterial spin label MRI with Xenon contrast agent to assess collateral blood flow.
  Interventions: Drug: Xenon contrast agent; Device: Magnetic Resonance Imaging
- Diagnosis unspecified (Experimental): Approximately 60 participants with diagnosis unspecified will be enrolled, and will receive arterial spin label MRI with Xenon contrast agent to assess collateral blood flow.
  Interventions: Drug: Xenon contrast agent; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Xenon contrast agent
  Other Names: XeMED contrast agent
Device: Magnetic Resonance Imaging — Arterial spin label sequence for the purpose of measuring collateral flow

SUMMARY:
Quantifying Collateral Perfusion in Cerebrovascular Disease-Moyamoya disease and stroke patients

DETAILED DESCRIPTION:
In the early hours following large vessel occlusion, the ultimate severity of the stroke is largely determined by the ability of collateral flow networks to supply blood to ischemic tissue via circuitous routes that bypass the proximal clot. Robust collateral flow can improve response to thrombolytic therapy and decrease the risk of intracranial hemorrhage. Despite their central importance, collaterals during acute stroke are poorly understood, largely because assessment has required an invasive imaging test, cerebral angiography. This proposal assesses whether a noncontrast MRI perfusion technique, called arterial spin labeling (ASL), can yield important information about collateral flow.

ELIGIBILITY:
Inclusion Criteria:

Moyamoya Patient Inclusion Criteria:

* Men and non-pregnant women, at least 21 years of age.
* Outpatients seen at the Stanford Neurosurgery and Neurology Departments.
* Ability to comply with all studies.
* Inclusion of Moyamoya patients with Sulfa allergies.
* Patients diagnosed with or suspected to have Moyamoya disease.

Stroke Patient Inclusion Criteria:

* Men and non-pregnant women, at least 21 years of age.
* Patients admitted to the inpatient Stanford Stroke Service for stroke-like symptoms, less than 24 hours from last time seen normal.
* Ability to comply with all studies.

Clinical Patient Acetazolamide MRI Inclusion Criteria:

* Men and non-pregnant women, at least 21 years of age.
* Patients admitted to the inpatient Stanford Stroke Service or Neurosurgical -Service for symptoms compatible with cerebrovascular disease.
* Ability to comply with all studies.

Normal Subject Inclusion Criteria:

* Ability to comply with the MRI study.

Exclusion Criteria:

* Level of consciousness score of 2 or greater as defined by the NIH stroke scale.
* Symptoms likely related to psychoactive drugs or patients with symptoms related to an active inflammatory disease such as AIDS, meningitis, or cerebritis.
* Psychiatric or substance abuse disorder or dementia that interferes with evaluation or interpretation of the neurologic and mental assessment of these patients.
* Informed consent cannot be obtained either from the patient or legal representative.
* Severe coexisting or terminal systemic disease that limits life expectancy or that may interfere with the conduct of the study.
* Symptoms related to an alternative diagnosis such as seizures or migraine.
* Patients receiving any thrombolytic agent or receiving acute stroke investigational drug therapies during the 30-day study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Zaharchuk, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was closed prior to any enrollment in the acute stroke, healthy participant, and diagnosis unspecified groups, so results are presented for the Moyamoya group only.
Groups:
- Moyamoya: Participants with Moyamoya disease received arterial spin label magnetic resonance imaging (MRI) with xenon contrast agent.
Period: Overall Study
Arm/Group | Moyamoya
Started | 126
Completed | 126
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Moyamoya: Participants with Moyamoya disease received arterial spin label MRI with xenon contrast agent.
Arm/Group | Moyamoya
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 37
Region of Enrollment [Number; unit: participants]
  United States | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Regions With Collateral Versus Antegrade Blood Flow (Sensitivity) Correctly Identified Using MRI With Xenon Contrast Agent (Specificity)
Description: Sensitivity and specificity for MRI-based ASL measure of presence of collaterals was measured using digital subtraction angiography as a gold standard. Measurements were for 20 regions per patient were scored as either positive or negative for collateral flow. A positive value (results) means the region is supplied by collateral flow. Negative means the region is supplied by antegrade (normal) flow. Sensitivity measures the proportion of positives that are correctly identified as such. Specificity measures the proportion of negatives that are correctly identified as such.
Time Frame: performed one time within 1 week prior to surgery
Population: One participant did not undergo MRI and was not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of regions
Units Other Than Participants: Cerebral regions
Arm/Group | Moyamoya
Number analyzed (Participants) | 125
Number analyzed (Cerebral regions) | 2500
percentage of regions
  Sensitivity | 81.7 [79.3 to 84.0]
  Specificity | 88.9 [86.6 to 90.8]

ADVERSE EVENTS:
Time Frame: 2 days
Description: Observed subjects for allergic reactions or other adverse events.
Arm/Group | Moyamoya
Serious Adverse Events (participants affected / at risk) | 0/126
Other Adverse Events (participants affected / at risk) | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes